CLINICAL TRIAL: NCT03731910
Title: Short Term Magnetic Resonance Imaging (MRI) for Treatment Response Evaluation and Prognosis Prediction in Patients With Hepatocellular Carcinoma (HCC) Treated With Transarterial Radioembolization (TARE)
Brief Title: Short-term MRI for Treatment Response Evaluation/Prediction of HCC Treated With TARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dongkook Lifesicence (Unknown)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNUH-1807-149-957
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCC group (Experimental): Participants who are scheduled for TARE for HCC treatment. They undergo MRI three times- before, 1- and 2-week after TARE.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — liver MRI using standard dose of extracellular agent. It includes dynamic contrast-enhanced MRI and diffusion weighted image.
  Other Names: magnetic resonance imaging

SUMMARY:
This study aims to investigate the value of early change at MRI in HCC treated with TARE, for evaluation/prediction of treatment response and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate or locally advanced HCC according to Hong Kong Liver Cancer guideline
* Scheduled for transarterial radioembolization (TARE)
* sign informed consent

Exclusion Criteria:

* Any absolute or relative contra-indication of contrast-enhanced MRI
* History of other local treatment before TARE in 3 weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment response mRECIST | 1 month after last MRI
  treatment response using mRECIST

SECONDARY OUTCOMES:
Tumor diffusion | 1 months after last MRI
  measured with diffusion-weighted image sequence
Tumor perfusion | 1 months after last MRI
  measured with dynamic contrast-enhanced imaging
Treatment response LI-RADS | 1 months after last MRI
  treatment response using LI-RADSv 2018 treatment response category
Treatment response volumetric | 1 months after last MRI
  treatment response using volumetric response criteria
Time to Progression | 24 months after TARE
  Time until to definite progression on follow-up images

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No